CLINICAL TRIAL: NCT05326893
Title: Preventive Effect of Femoral Nerve Neurodynamic Mobilization Against Maximal Eccentric Exercise-induced Muscle Damage of the Knee Extensors: a Randomized, Single-blinded, Sham-Controlled Study
Brief Title: The Preventive Effects of Neurodynamic Mobilisation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uğur Sözlü (Other)
Collaborators: Gazi University (Other)
Responsible Party: Sponsor-Investigator, Uğur Sözlü, Principal Investigator, Gazi University
Organization: Gazi University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 02.10.2019 / 270
Record Dates: First submitted 2022-03-29; First posted 2022-04-14 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Delayed Onset Muscle Soreness
Keywords: Delayed onset muscle soreness; Neurodynamic mobilization; Muscle damage; Inflammation; Pain
MeSH Terms: conditions — Inflammation; Pain

STUDY DESIGN:
Intervention Model Description: The study was conducted as a randomized, single-blind, sham-controlled clinical trial.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Femoral nerve neurodynamic mobilization group
  T1: Baseline measurements were made and blood samples were taken for biochemical analysis.
  NM and placebo NM techniques were applied for three weeks, three times a week, and totaling nine visits. At the end of the third week, it was waited 3 days to eliminate the acute effect of NM.
  T2: Baseline measurements and blood samples were repeated a second time.
  The protocol for establishing the DOMS was applied on the same day.
  T3: Following the protocol for inducing the DOMS, the baseline measurements were repeated for the third time without any interruption, and the blood sample was taken.
  T4-T5-T6: The first measurements and blood sample collections were repeated for the fourth, fifth and sixth times, respectively, 24h, 48h, 72h after the DOMS protocol.
  Interventions: Other: Femoral nerve neurodynamic mobilization
- Placebo Group (Placebo Comparator): Femoral nerve placebo neurodynamic mobilization group
  T1: Baseline measurements were made and blood samples were taken for biochemical analysis.
  NM and placebo NM techniques were applied for three weeks, three times a week, and totaling nine visits. At the end of the third week, it was waited 3 days to eliminate the acute effect of NM.
  T2: Baseline measurements and blood samples were repeated a second time.
  The protocol for establishing the DOMS was applied on the same day.
  T3: Following the protocol for inducing the DOMS, the baseline measurements were repeated for the third time without any interruption, and the blood sample was taken.
  T4-T5-T6: The first measurements and blood sample collections were repeated for the fourth, fifth and sixth times, respectively, 24h, 48h, 72h after the DOMS protocol.
  Interventions: Other: Femoral nerve placebo neurodynamic mobilization

INTERVENTIONS:
Other: Femoral nerve neurodynamic mobilization — The mobilization was carried out with the patient lying on the non-dominant side in a total flexion position, and the therapist performed the hip extension movement with the knee joint kept in flexion till the patient felt soreness or pain. This position was held for three seconds and then released. This tensioning maneuver was repeated in three sets of ten repetitions at each session and an interval of 2 min between series were performed. A total of nine sessions were performed within three weeks.
  Arms: Study Group
Other: Femoral nerve placebo neurodynamic mobilization — The individual was asked to lie on his non-dominant side and keep his head in the midline. In this position, while the pelvis was stabilized, the upper leg, which was in full knee extension, was grasped and the hip was abducted for 3 seconds. This maneuver was repeated in three sets of ten repetitions at each session and an interval of 2 min between series were performed. A total of nine sessions were performed within three weeks.
  Arms: Placebo Group

SUMMARY:
In the study, 34 healthy sedentary male volunteers were randomly divided into two groups as NM (n = 17) and SHAM-NM (n = 17). After the initial evaluation of the individuals, femoral nerve NM and placebo NM techniques were administered three sets a day with ten repetitions for three days a week for three weeks. Three days after the end of the applications, the second evaluations were made and the DOMS creation protocol for the quadriceps femoris (QF) muscle was initiated. In order to trigger DOMS in individuals, 30 sets and 10 repetitions of eccentric knee extension (35°-95° flexion angles, 30°/sec speed) were performed on the dominant lower extremity with an isokinetic dynamometer. Baseline evaluations were repeated immediately after the DOMS protocol, and at hours 24, 48, and 72. During evaluations, muscle damage (serum creatine kinase (CK), lactate dehydrogenase (LDH), and inflammation (interleukin-6 (IL-6), tumor necrosis factor-alpha) biomarkers, pain (activity), pressure pain threshold, and performance (one-leg jump, vertical jump) parameters were measured.

DETAILED DESCRIPTION:
The aim of this study was to investigate the effects of neurodynamic mobilization (NM) technique on muscle damage and inflammation biomarkers, and pain, pressure pain threshold, and functional status in delayed onset muscle soreness (DOMS). In the study, 34 healthy sedentary male volunteers were randomly divided into two groups as NM (n = 17) and SHAM-NM (n = 17). After the initial evaluation of the individuals, femoral nerve NM and placebo NM techniques were administered three sets a day with ten repetitions for three days a week for three weeks. Three days after the end of the applications, the second evaluations were made and the DOMS creation protocol for the quadriceps femoris (QF) muscle was initiated. In order to trigger DOMS in individuals, 30 sets and 10 repetitions of eccentric knee extension (35°-95° flexion angles, 30°/sec speed) were performed on the dominant lower extremity with an isokinetic dynamometer. Baseline evaluations were repeated immediately after the DOMS protocol, and at hours 24, 48, and 72. During evaluations, muscle damage (serum creatine kinase (CK), lactate dehydrogenase (LDH), and inflammation (interleukin-6 (IL-6), tumor necrosis factor-alpha) biomarkers, pain (activity), pressure pain threshold, and performance (one-leg jump, vertical jump) parameters were measured.

ELIGIBILITY:
Inclusion Criteria:

* Being in the age range of 20-32 years.
* Being male (Because gender difference in the magnitude of eccentric exercise-induced muscle damage might exist as shown in previous studies, only men were recruited in the present study.)
* Being inactive according to activity guidelines published by the American College of Sports Medicine (less than 30 minutes of moderate physical activity as five times a week).

Exclusion Criteria:

* Absence of DOMS symptoms,
* History of vascular disease,
* Recent injury or surgery to their lower extremity,
* Neurological impairments and regular use of pain and inflammation medications.

Ages: 18 Years to 32 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Muscle Soreness at 4 weeks | up to 4 weeks
  Muscle soreness was assessed using a 100 mm visual analog scale (0 = no soreness, 10 = excruciatingly painful). Each subject walked down 10 steps of stairs and asked to indicate the soreness level on the line. The marked point was measured with a ruler and recorded in millimeters.
Change from Baseline Muscle damage marker (Creatine kinase (U/L)) at 4 weeks | up to 4 weeks
  Creatine kinase (U/L) was assessed using an enzyme-linked immunoassay as per the manufacturer's protocol (Beckman Coulter, Inc., CA, U.S.A.).
Change from Baseline Muscle damage marker (Laktat dehidrogenaz (U/L)) at 4 weeks | up to 4 weeks
  Lactate dehydrogenase (U/L) was assessed using an enzyme-linked immunoassay as per the manufacturer's protocol (Beckman Coulter, Inc., CA, U.S.A.).
Change from Baseline Inflammatory stress marker (Tumor necrosis factor-alfa ((pg/ml)) at 4 weeks | up to 4 weeks
  Tumor necrosis factor-alfa (pg/ml), was assessed using a sandwich enzyme linked immunoassay test as per the manufacturer's protocol.
Change from Baseline Inflammatory stress marker (Human interleukin-6 (pg/ml)) at 4 weeks | up to 4 weeks
  Human interleukin-6 ((pg/ml)), was assessed using a sandwich enzyme linked immunoassay test as per the manufacturer's protocol.
Change from Baseline Pressure Pain Threshold (N/cm2) at 4 weeks | up to 4 weeks
  The pressure pain threshold ((N/cm2) ) was measured using a digital pressure algometer (JTECH Medical Industries, Salt Lake City, US) at the midpoint of quadriceps femoris muscle and the other at 5 cm above the superior pole of the patella (representing the musculotendinous junction). The average value of three trials was used in the analysis. PPT measurements were found to have acceptable intra and inter-observer reliability (ICC 0.7).
Change from Baseline One leg hop test (cm) at 4 weeks | up to 4 weeks
  In the one leg hop test (cm), participants required to stand on one leg to be tested, to jump off and to land on that leg without losing balance. Three hops (with 60 sec rest between hops) were performed and the distance hopped was measured with a standard tape measure. Mean value of distance was recorded as centimeter.

CONTACTS AND LOCATIONS:
Overall Officials: Selda Başar, Phd, Study Chair — Gazi University
Locations (1):
- Gazi University, Ankara, Beşevler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sozlu U, Basar S, Semsi R, Akaras E, Sepici Dincel A. Preventive effect of the neurodynamic mobilization technique on delayed onset of muscle soreness: a randomized, single-blinded, placebo-controlled study. BMC Musculoskelet Disord. 2025 May 10;26(1):464. doi: 10.1186/s12891-025-08723-8. PMID 40349018